CLINICAL TRIAL: NCT06290908
Title: Robot-assisted Percutaneous Endoscopic Posterior/Transforaminal Lumbar Interbody Fusion for Lumbar Spinal Stenosis With Instability
Brief Title: RPE-P/TLIF for Lumbar Spinal Stenosis With Instability
Status: Completed | Type: Observational
Sponsor: Wen-xi Sun (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Wen-xi Sun, Clinical Professor, Guangzhou University of Chinese Medicine
Organization: Guangzhou University of Chinese Medicine (Other)
Other Study IDs: TF2018-001-01
Record Dates: First submitted 2024-02-20; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RPE-P/TLIF: The clinical manifestation is intermittent claudication accompanied by lower back pain. Patients with lumbar spinal canal stenosis indicated by MRI and/or CT, and instability of the responsible segment of the lumbar spine shown by X-ray in the over extension and over flexion position, with severe symptoms that affect daily life and work, and poor conservative treatment effect, should undergo RPE-P/TLIF single or double segment surgical treatment.
  Interventions: Procedure: RPE-P/TLIF

INTERVENTIONS:
Procedure: RPE-P/TLIF — patients with lumbar spinal stenosis and instability who met the inclusion and exclusion criteria were treated with RPE-P/TLIF

SUMMARY:
Objective To analyze the effectiveness and safety of robot-assisted percutaneous endoscopic posterior/transforaminal lumbar interbody fusion (RPE-P/TLIF) in the treatment of lumbar spinal stenosis with instability. Methods A single-center prospective study from September 2018 to April 2022, patients with lumbar spinal stenosis and instability who met the inclusion and exclusion criteria were treated with RPE-P/TLIF. Pain visual analog scale (VAS) was used to evaluate the degree of low back pain and lower limb pain before operation, 1 month, 6 months, 1 year after operation and at the final follow-up, and the Oswestry disability index (ODI) was used to evaluate the degree of lumbar spinal function. At the last follow-up, MacNab criteria were used to evaluate the clinical efficacy. Imaging evaluation included the measurement of intervertebral space height, lumbar physiological curvature, fusion rate and pedicle screw accuracy by preoperative and lateral X-ray films.

ELIGIBILITY:
Inclusion Criteria:

Patients who present with intermittent claudication accompanied by lower back pain, lumbar spine MRI and/or CT findings of lumbar spinal stenosis, and X-ray images of over extension and over flexion indicating instability of the responsible segment of the lumbar spine, have severe symptoms that affect daily life and work, and have poor conservative treatment results. Therefore, RPE-P/TLIF single segment or double segment surgical treatment is recommended.

Exclusion Criteria:

(1) Simple lumbar spinal stenosis without responsible segment instability; (2) Long segment (3 or more) spinal stenosis with lumbar instability; (3) Patients with major internal medicine underlying diseases who cannot tolerate surgery; (4) Individuals with comorbid mental disorders or Alzheimer's disease who are unable to cooperate with relevant scale filling and subsequent follow-up; (5) Age<18 years old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included patients with clinical manifestations of intermittent claudication accompanied by lower back pain, lumbar spine MRI and/or CT findings of lumbar spinal stenosis, and X-ray images of over extension and over flexion indicating responsible segment lumbar instability. Symptoms were severe, affecting daily life and work, and conservative treatment was ineffective. RPE-P/TLIF single or double segment surgery was performed.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Pain visual analog scale (VAS) | Before surgery, 1 month after surgery, 6 months after surgery, 1 year after surgery, and 4 years after surgery
  Pain assessment, assessing lower back pain and lower limb pain.

SECONDARY OUTCOMES:
Oswestry disability index (ODI) | Before surgery, 1 month after surgery, 6 months after surgery, 1 year after surgery, and 4 years after surgery
  Evaluate neurological function
MacNab criteria | Before surgery, 1 month after surgery, 6 months after surgery, 1 year after surgery, and 4 years after surgery
  The overall efficacy rate was evaluated using the modified MacNab criteria, which were divided into four levels: excellent, good, fair, and poor. Among them, excellent was the complete disappearance of symptoms and the restoration of normal life; Liangwei still has mild symptoms and mild activity restriction, but has no impact on life and work; May still have obvious symptoms, limited activities, and affect normal life and work; Poor symptoms do not improve, activities do not improve, and even worsen.
intervertebral space height | Before surgery, 1 month after surgery, 6 months after surgery, 1 year after surgery, and 4 years after surgery
  Imaging evaluation indicators:
lumbar physiological curvature | Before surgery, 1 month after surgery, 6 months after surgery, 1 year after surgery, and 4 years after surgery
  Imaging evaluation indicators:
fusion rate | Before surgery, 1 month after surgery, 6 months after surgery, 1 year after surgery, and 4 years after surgery
  Imaging evaluation indicators:
pedicle screw accuracy | Before surgery, 1 month after surgery, 6 months after surgery, 1 year after surgery, and 4 years after surgery
  Imaging evaluation indicators:

CONTACTS AND LOCATIONS:
Overall Officials: Yong-peng Lin, dr, Study Chair — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided
We are considering sharing our IPD after the data statistics are completed.